CLINICAL TRIAL: NCT06584838
Title: Primary ACL Reconstruction in Patient Over 40 Years: Allograft Versus Autograft, a Prospective Matched Paired Comparison
Brief Title: Primary ACL Reconstruction in Patient Over 40 Years: Allograft Versus Autograft
Status: Not yet recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Professor Giacomo Placella, Professor, IRCCS Ospedale San Raffaele
Other Study IDs: ALVSAT
Record Dates: First submitted 2024-07-29; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: ACL; ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Allograft: Patients aged ≥ 40 y.o. that underwent ACL reconstruction using allograft tendons
  Interventions: Procedure: ACL reconstruction
- Autograft: Patients aged ≥ 40 y.o. that underwent ACL reconstruction using autograft tendons
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — Patients that underwent ACL reconstruction using either allograft or autograft tendons, at least 2 years of follow-up, gender male and female, no comorbidities

SUMMARY:
The aim of this study is to investigate the differences in graft failure between patients that underwent ACL reconstruction using allograft tendons and patients that underwent ACL reconstruction using autograft tendons in patients older than 40 y.o. and after at least 2 years of follow-up. The hypothesis of the study is that there will be a difference in graft failure and patient reported functional outcomes between allograft and autograft ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male and female patients of fertile age can be recruited
* Patients aged 40 years old and above, and 2 years minimum of follow-up
* Patients that underwent primary ACL reconstruction with allograft an autograft tendons

Exclusion Criteria:

* Multiligamentous lesion
* Meniscal tear leading to subtotal or total meniscectomy or meniscal graft
* Indication for major cartilage restoration or resurfacing
* Ipsilateral knee fractures
* History of ligament injury
* Concomitant extracapsular procedures
* Ipsilateral or contralateral knee surgeries

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that underwent ACL reconstruction using either allograft or autograft tendons, at least 2 years of follow-up, gender male and female, no comorbidities.
  Group 1 are patients aged ≥ 40 y.o. that underwent ACL reconstruction using allograft tendons.
  Group 2 are patients aged ≥ 40 y.o. that underwent ACL reconstruction using autograft tendons.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
To compare the difference in graft failure between allograft vs autograft ACL reconstruction | from 2 years after surgical procedure
  Clinical evaluation measuring the percentage in graft failure between allograft and autograft ACL reconstruction

SECONDARY OUTCOMES:
To assess the difference in patient reported outcome between allograft vs autograft ACL reconstruction | from 2 years after surgical procedure
  Clinical evaluation collecting Tegner Lysholm Score (max, 100 - min. 0) (100 = no disability; 0= maximum siability)
To assess the difference in patient reported outcome between allograft vs autograft ACL reconstruction | from 2 years after surgical procedure
  Clinical evaluation collecting the Visual Analogue Scale for Pain (VAS) (min.0 - max. 10) (0= no pain; 100 maximum pain)
To assess the difference in patient reported outcome between allograft vs autograft ACL reconstruction | from 2 years after surgical procedure
  Clinical evaluation collecting the International Knee Document Comitee Score (IKDC) (min. 0 - max. 100) (0= lowest level of function; 100= highest level of fuction)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barrett G, Stokes D, White M. Anterior cruciate ligament reconstruction in patients older than 40 years: allograft versus autograft patellar tendon. Am J Sports Med. 2005 Oct;33(10):1505-12. doi: 10.1177/0363546504274202. Epub 2005 Jul 11. PMID 16009990
- [Background] Seng K, Appleby D, Lubowitz JH. Operative versus nonoperative treatment of anterior cruciate ligament rupture in patients aged 40 years or older: an expected-value decision analysis. Arthroscopy. 2008 Aug;24(8):914-20. doi: 10.1016/j.arthro.2008.01.021. Epub 2008 Apr 18. PMID 18657740
- [Background] Kuechle DK, Pearson SE, Beach WR, Freeman EL, Pawlowski DF, Whipple TL, Caspari Dagger RB, Meyers JF. Allograft anterior cruciate ligament reconstruction in patients over 40 years of age. Arthroscopy. 2002 Oct;18(8):845-53. doi: 10.1053/jars.2002.36140. PMID 12368781
- [Background] Budny J, Fox J, Rauh M, Fineberg M. Emerging Trends in Anterior Cruciate Ligament Reconstruction. J Knee Surg. 2017 Jan;30(1):63-69. doi: 10.1055/s-0036-1579788. Epub 2016 Mar 28. PMID 27018510
- [Background] Tibor L, Chan PH, Funahashi TT, Wyatt R, Maletis GB, Inacio MC. Surgical Technique Trends in Primary ACL Reconstruction from 2007 to 2014. J Bone Joint Surg Am. 2016 Jul 6;98(13):1079-89. doi: 10.2106/JBJS.15.00881. PMID 27385681
- [Background] Salminen M, Kraeutler MJ, Freedman KB, Tucker BS, Salvo JP, Ciccotti MG, Cohen SB. Choosing a Graft for Anterior Cruciate Ligament Reconstruction: Surgeon Influence Reigns Supreme. Am J Orthop (Belle Mead NJ). 2016 May-Jun;45(4):E192-7. PMID 27327925
- [Background] Joyce CD, Randall KL, Mariscalco MW, Magnussen RA, Flanigan DC. Bone-Patellar Tendon-Bone Versus Soft-Tissue Allograft for Anterior Cruciate Ligament Reconstruction: A Systematic Review. Arthroscopy. 2016 Feb;32(2):394-402. doi: 10.1016/j.arthro.2015.08.003. Epub 2015 Sep 28. PMID 26427630
- [Background] Kaeding CC, Pedroza AD, Reinke EK, Huston LJ; MOON Consortium; Spindler KP. Risk Factors and Predictors of Subsequent ACL Injury in Either Knee After ACL Reconstruction: Prospective Analysis of 2488 Primary ACL Reconstructions From the MOON Cohort. Am J Sports Med. 2015 Jul;43(7):1583-90. doi: 10.1177/0363546515578836. Epub 2015 Apr 21. PMID 25899429